CLINICAL TRIAL: NCT05580549
Title: Prevalence of Hazardous Alcohol Use in a Population With Hypertension in Primary Care Detected With PEth and AUDIT - Observational Cross-sectional Study
Brief Title: Prevalence of Hazardous Alcohol Use in a Population With Hypertension in Primary Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other); Forte (Industry); Sophiahemmet University (Other)
Responsible Party: Sponsor
Other Study IDs: SLSO2022-0143
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Hypertension; Alcohol Drinking; Alcohol Use, Unspecified
Keywords: Phosphatidylethanol; Alcohol Use Disorders Identification Test (AUDIT); Primary Health Care; Health promotion
MeSH Terms: conditions — Hypertension; Alcohol Drinking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood fats (P-Cholesterol, P-HDL, P-LDL, fP-Triglycerides) Glucose (fP-glucose) Blood status (B-Hemoglobin, B-EVF, B-MCV, B-MCH, B-MCHC, B-Leucocytes, B-Thrombocytes Kidney function (P-Creatinine, P-Potassium, U-Albumin/Creatinine, Pt-eGFR) Phosphatidylethanol ( B-PEth 16:0/18:1)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Essential Hypertension: A representative sample of adult patients, with hypertension (ICD-10 diagnose code I10.9) from 2-3 PHCC in Stockholm Region, Sweden. Age 30-85 years old.
  Interventions: Diagnostic Test: Alcohol biomarker Phosphatidylethanol (PEth)

INTERVENTIONS:
Diagnostic Test: Alcohol biomarker Phosphatidylethanol (PEth) — The prevalence of hazardous alcohol use will be mapped through the biomarker PEth and the questionnaire AUDIT.
  Other Names: Alcohol Use Disorders Identification Test (AUDIT)

SUMMARY:
The goal of this observational cross-sectional study is to map the prevalence of hazardous alcohol use in 270 adult patients with hypertension in Primary Health Care (PHC). The main question it aims to answer is: What is the prevalence of hazardous alcohol use in a population with hypertension in primary care detected with PEth and AUDIT, analysed in relation to patients with controlled, uncontrolled and treatment resistant hypertension? Participants will, in conjunction with annual control of hypertension with a General Practitioner (GP) at their Primary Health Care Centre (PHCC), visit a study nurse. The study nurse will collect following data: • Physical measurements• Lifestyle habits• Quality of life and demographic data • Drugs for hypertension and comorbidity • Laboratory tests including Phosphatidylethanol (PEth).

DETAILED DESCRIPTION:
Hypertension, tobacco smoking, and alcohol use are the three leading risk factors for global disease burden. Treatment of hypertensive disease is important for the prevention of atherosclerotic disease, atrial fibrillation, heart failure, stroke, and dementia. In Sweden 27 % of adults have hypertension and a majority are treated in PHC but only 37 % reach target blood pressure. Alcohol can be one factor behind the low number of goal completion of blood pressure level.

Prevalence of hazardous alcohol use in Sweden is between 10-30 % in adults. Alcohol has an important role for over 200 diagnoses. There is a causal and dose dependent relationship between blood pressure levels and regular alcohol intake. Previous studies have reported hypertension to be attributable to alcohol in a wide range, depending on for example population, sex, and cultural context. But studies about the prevalence of hazardous alcohol use in patients with hypertension is few or even lacking.

General Practitioners (GPs) miss to identify a majority (60-70%) of patients with hazardous alcohol use even though guidelines on hypertension include risk stratification and detection of harmful lifestyle and the fact that general practitioners find it important to talk about alcohol with their patients.

Alcohol Use Disorders Identification Test (AUDIT) is a validated screening test for hazardous and harmful use in PHC setting, although concerns have been raised to its sensitivity. GPs experience that patient underestimate their consumption and that AUDIT does not meet the requirements to be a useful tool to detect hazardous alcohol use and AUDIT is seldomly used in PHC.

The alcohol biomarker Phosphatidylethanol (PEth) has high sensitivity and specificity to detect alcohol use. PEth can detect chronic heavy consumption. PEth is one of the newest alcohol biomarkers, but despite promising characteristics of PEth it is not routinely applied in clinical practice. PEth is used in a variety of settings like addiction care, emergency rooms, treatment of HIV-patients and patients with liver disease. PEth has started to be used in PHC but few studies on the use of biomarkers for alcohol consumption have been carried out in PHC.

The Swedish National Board of Health and Welfare has presented methods to use for supporting patients to change hazardous alcohol use. First the GPs need to identify if the patient has hazardous alcohol use. To our knowledge studies on whether PEth is a useful tool to detect hazardous use in patients with hypertension, in a primary health care context, is scarce or missing.

Study design

Based on that 12% of the hypertensive patients is related to alcohol intake and a presumed prevalence of hazardous drinking of 15 % the required sample size, given an effect size of 21%, significance level 5%, and power of 80% using contingency tables with 2 degrees of freedom, the study will require 270 patients with an included 10 % to compensate for missing values.

To perform an effective recruitment of patients we will invite patients from three well-functioning PHCCs with approximately 15.000 listed patients. Criteria for well-functioning is stable management and staff, routines for handling hypertension as well as unhealthy life-style habits and ability to offer locals for the project. By using the tool Medrave4 all patients 30-85 years old with hypertension (ICD-10 diagnose code I10.9) will be extracted from the PHCCs. The patients will be stratified to three groups of hypertension: •Controlled (blood pressure < 140/90), •Uncontrolled (blood pressure ≥ 140/90) and, •Treatment resistant hypertension (≥ 140/90 with three or more drugs against hypertension). Strata groups will be randomised, and the patients will be invited top to bottom. Recruitment will stop when 30 patients from each group has been included.

The PHCCs operations manager invites patients by letter. Patients have the opportunity to register their interest in participating in the study by letter or phone. Patients can also notify that they do not wish to be contacted. After 2-3 weeks the study nurse calls the patients and ask if they want to participate. The study nurse makes an initial assessment of the inclusion and exclusion criteria over the phone.

At the visit with the study nurse the final assessment of inclusion and exclusion criteria will be made. Finally the patients will be included after written informed consent. At the visit following data will be collected and stored at the digital platform REDCap:• Physical measurements (Blood pressure, pulse, weight, height, and waist measurement) • Lifestyle habits ( Alcohol, tobacco, food, and physical activity) • Quality of life (EQ-5D-5L) •Comorbidity with relevance to hypertension (Diabetes type 1 or 2, atrial fibrillation, angina pectoris, heart failure, myocardial infarction, stroke, and Transient ischemic attack) • Socioeconomic data (year of birth, gender, education, employment, occupation, people in the household) • Drugs for hypertension (Beta blockers, Calcium blockers, Thiazides, ACE inhibitors, ARB blockers, and Potassium-sparing diuretic) • Blood- and urine tests for hypertension and Phosphatidylethanol (PEth).

Patients will then visit their GP for an usual annual control of hypertension. The patients will receive results of blood tests and if needed adjustment of treatment will be done. Study nurse and GPs will talk about life style factors, including alcohol, with the patient. If hazardous alcohol use they will give short advice and offer more support if the patient needs and wants it. Before the start of the study GPs from the PHCCs will attend a short education of how to interpret PEth and AUDIT.

Detection of hazardous alcohol use, by the two methods PEth and AUDIT, will be described in the three strata (controlled, uncontrolled and treatment resistant hypertension) of the whole cohort. We will adjust for possible confounders (lifestyle factors, socio-economic data and patients' perceived health). We will relate our calculations to established risk stratification models for cardiovascular disease. All patients with hypertension and the drop-out population will be analysed according to what is ethically possible. Usual statistical presentation methods based on the scale level of collected data and other properties will be used.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension ICD-10 code I10.9.
* Age 30-85 years.

Exclusion Criteria:

* Not able to come to the primary health care centre
* Not understanding swedish
* Not speaking swedish
* Severe disease
* Dementia
* Serious mental illness

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From 2-3 PHCCs, in Stockholm region in Sweden, we will find patients with the extraction tool Medrave4. Patients with hypertension from the last two years will be extracted and the criteria for inclusion will be applied. A stratified and random sample will be created of three different groups of hypertension: Controlled, Uncontrolled and, Treatment resistant hypertension.
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Hazardous alcohol use | baseline
  Measured PEth-value. Defined as > 0,3 µmol/L on PEth.
Hazardous alcohol use | Baseline
  Selfreported values. Defined as 6-13 points for women and 8-15 points for men on Alcohol Use Disorders Identification Test (AUDIT).

CONTACTS AND LOCATIONS:
Overall Officials: Lena Lund, PhD, Principal Investigator — Region Stockholm
Locations (1):
- Region Stockholm, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lim SS, Vos T, Flaxman AD, Danaei G, Shibuya K, Adair-Rohani H, Amann M, Anderson HR, Andrews KG, Aryee M, Atkinson C, Bacchus LJ, Bahalim AN, Balakrishnan K, Balmes J, Barker-Collo S, Baxter A, Bell ML, Blore JD, Blyth F, Bonner C, Borges G, Bourne R, Boussinesq M, Brauer M, Brooks P, Bruce NG, Brunekreef B, Bryan-Hancock C, Bucello C, Buchbinder R, Bull F, Burnett RT, Byers TE, Calabria B, Carapetis J, Carnahan E, Chafe Z, Charlson F, Chen H, Chen JS, Cheng AT, Child JC, Cohen A, Colson KE, Cowie BC, Darby S, Darling S, Davis A, Degenhardt L, Dentener F, Des Jarlais DC, Devries K, Dherani M, Ding EL, Dorsey ER, Driscoll T, Edmond K, Ali SE, Engell RE, Erwin PJ, Fahimi S, Falder G, Farzadfar F, Ferrari A, Finucane MM, Flaxman S, Fowkes FG, Freedman G, Freeman MK, Gakidou E, Ghosh S, Giovannucci E, Gmel G, Graham K, Grainger R, Grant B, Gunnell D, Gutierrez HR, Hall W, Hoek HW, Hogan A, Hosgood HD 3rd, Hoy D, Hu H, Hubbell BJ, Hutchings SJ, Ibeanusi SE, Jacklyn GL, Jasrasaria R, Jonas JB, Kan H, Kanis JA, Kassebaum N, Kawakami N, Khang YH, Khatibzadeh S, Khoo JP, Kok C, Laden F, Lalloo R, Lan Q, Lathlean T, Leasher JL, Leigh J, Li Y, Lin JK, Lipshultz SE, London S, Lozano R, Lu Y, Mak J, Malekzadeh R, Mallinger L, Marcenes W, March L, Marks R, Martin R, McGale P, McGrath J, Mehta S, Mensah GA, Merriman TR, Micha R, Michaud C, Mishra V, Mohd Hanafiah K, Mokdad AA, Morawska L, Mozaffarian D, Murphy T, Naghavi M, Neal B, Nelson PK, Nolla JM, Norman R, Olives C, Omer SB, Orchard J, Osborne R, Ostro B, Page A, Pandey KD, Parry CD, Passmore E, Patra J, Pearce N, Pelizzari PM, Petzold M, Phillips MR, Pope D, Pope CA 3rd, Powles J, Rao M, Razavi H, Rehfuess EA, Rehm JT, Ritz B, Rivara FP, Roberts T, Robinson C, Rodriguez-Portales JA, Romieu I, Room R, Rosenfeld LC, Roy A, Rushton L, Salomon JA, Sampson U, Sanchez-Riera L, Sanman E, Sapkota A, Seedat S, Shi P, Shield K, Shivakoti R, Singh GM, Sleet DA, Smith E, Smith KR, Stapelberg NJ, Steenland K, Stockl H, Stovner LJ, Straif K, Straney L, Thurston GD, Tran JH, Van Dingenen R, van Donkelaar A, Veerman JL, Vijayakumar L, Weintraub R, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams W, Wilson N, Woolf AD, Yip P, Zielinski JM, Lopez AD, Murray CJ, Ezzati M, AlMazroa MA, Memish ZA. A comparative risk assessment of burden of disease and injury attributable to 67 risk factors and risk factor clusters in 21 regions, 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2224-60. doi: 10.1016/S0140-6736(12)61766-8. PMID 23245609
- [Background] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; ESC Scientific Document Group. 2018 ESC/ESH Guidelines for the management of arterial hypertension. Eur Heart J. 2018 Sep 1;39(33):3021-3104. doi: 10.1093/eurheartj/ehy339. No abstract available. PMID 30165516
- [Background] Holmquist C, Hasselstrom J, Bengtsson Bostrom K, Manhem K, Wettermark B, Hjerpe P, Kahan T. Improved treatment and control of hypertension in Swedish primary care: results from the Swedish primary care cardiovascular database. J Hypertens. 2017 Oct;35(10):2102-2108. doi: 10.1097/HJH.0000000000001429. PMID 28582282
- [Background] Rehm J, Gmel GE Sr, Gmel G, Hasan OSM, Imtiaz S, Popova S, Probst C, Roerecke M, Room R, Samokhvalov AV, Shield KD, Shuper PA. The relationship between different dimensions of alcohol use and the burden of disease-an update. Addiction. 2017 Jun;112(6):968-1001. doi: 10.1111/add.13757. Epub 2017 Feb 20. PMID 28220587
- [Background] Puddey IB, Mori TA, Barden AE, Beilin LJ. Alcohol and Hypertension-New Insights and Lingering Controversies. Curr Hypertens Rep. 2019 Sep 7;21(10):79. doi: 10.1007/s11906-019-0984-1. PMID 31494743
- [Background] Lang T, Degoulet P, Aime F, Devries C, Jacquinet-Salord MC, Fouriaud C. Relationship between alcohol consumption and hypertension prevalence and control in a French population. J Chronic Dis. 1987;40(7):713-20. doi: 10.1016/0021-9681(87)90108-1. PMID 3597673
- [Background] Marchi KC, Muniz JJ, Tirapelli CR. Hypertension and chronic ethanol consumption: What do we know after a century of study? World J Cardiol. 2014 May 26;6(5):283-94. doi: 10.4330/wjc.v6.i5.283. PMID 24944758
- [Background] Manthey J, Probst C, Hanschmidt F, Rehm J. Identification of smokers, drinkers and risky drinkers by general practitioners. Drug Alcohol Depend. 2015 Sep 1;154:93-9. doi: 10.1016/j.drugalcdep.2015.06.017. Epub 2015 Jun 22. PMID 26130336
- [Background] Hyland K, Hammarberg A, Andreasson S, Jirwe M. Treatment of alcohol dependence in Swedish primary care: perceptions among general practitioners. Scand J Prim Health Care. 2021 Jun;39(2):247-256. doi: 10.1080/02813432.2021.1922834. Epub 2021 Jun 21. PMID 34151724
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Higgins-Biddle JC, Babor TF. A review of the Alcohol Use Disorders Identification Test (AUDIT), AUDIT-C, and USAUDIT for screening in the United States: Past issues and future directions. Am J Drug Alcohol Abuse. 2018;44(6):578-586. doi: 10.1080/00952990.2018.1456545. Epub 2018 May 3. PMID 29723083
- [Background] Tam CW, Zwar N, Markham R. Australian general practitioner perceptions of the detection and screening of at-risk drinking, and the role of the AUDIT-C: a qualitative study. BMC Fam Pract. 2013 Aug 20;14:121. doi: 10.1186/1471-2296-14-121. PMID 23961835
- [Background] Nygaard P, Paschall MJ, Aasland OG, Lund KE. Use and barriers to use of screening and brief interventions for alcohol problems among Norwegian general practitioners. Alcohol Alcohol. 2010 Mar-Apr;45(2):207-12. doi: 10.1093/alcalc/agq002. Epub 2010 Jan 25. PMID 20100927
- [Background] Ulwelling W, Smith K. The PEth Blood Test in the Security Environment: What it is; Why it is Important; and Interpretative Guidelines. J Forensic Sci. 2018 Nov;63(6):1634-1640. doi: 10.1111/1556-4029.13874. Epub 2018 Jul 13. PMID 30005144
- [Background] Andresen-Streichert H, Muller A, Glahn A, Skopp G, Sterneck M. Alcohol Biomarkers in Clinical and Forensic Contexts. Dtsch Arztebl Int. 2018 May 4;115(18):309-315. doi: 10.3238/arztebl.2018.0309. PMID 29807559
- [Background] Viel G, Boscolo-Berto R, Cecchetto G, Fais P, Nalesso A, Ferrara SD. Phosphatidylethanol in blood as a marker of chronic alcohol use: a systematic review and meta-analysis. Int J Mol Sci. 2012 Nov 13;13(11):14788-812. doi: 10.3390/ijms131114788. PMID 23203094
- [Background] Aakeroy R, Skrastad RB, Helland A, Hilberg T, Aamo T, Dyrkorn R, Spigset O. [New biomarkers for assesing alcohol consumption]. Tidsskr Nor Laegeforen. 2016 Oct 25;136(19):1643-1647. doi: 10.4045/tidsskr.16.0056. eCollection 2016 Oct. Norwegian. PMID 27790892
- [Background] Topic A, Djukic M. Diagnostic characteristics and application of alcohol biomarkers. Clin Lab. 2013;59(3-4):233-45. PMID 23724610
- [Background] Miller PM, Anton RF. Biochemical alcohol screening in primary health care. Addict Behav. 2004 Sep;29(7):1427-37. doi: 10.1016/j.addbeh.2004.06.013. PMID 15345274
- [Background] Holte M, Holmen J. Program for data extraction in primary health records: a valid tool for knowledge production in general practice? BMC Res Notes. 2020 Jan 10;13(1):23. doi: 10.1186/s13104-020-4887-7. PMID 31924277
- [Background] Carlsson AC, Wandell P, Osby U, Zarrinkoub R, Wettermark B, Ljunggren G. High prevalence of diagnosis of diabetes, depression, anxiety, hypertension, asthma and COPD in the total population of Stockholm, Sweden - a challenge for public health. BMC Public Health. 2013 Jul 18;13:670. doi: 10.1186/1471-2458-13-670. PMID 23866784
- See also: The National Board of Health and Welfare 2018: National guidelines for disease prevention methods — https://www.socialstyrelsen.se/en/
- See also: The Central Association for Alcohol and Narcotic Information (CAN): Self-reported alcohol habits in Sweden 2004-2020. CAN report 204 — https://www.can.se/publikationer/sjalvrapporterade-alkoholvanor-i-sverige-2004-2020/